CLINICAL TRIAL: NCT05085392
Title: A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lauren Davis, Assistant Professor of Curriculum & Instruction, Montana State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MontanaSUYear3; P20GM104417 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Depression, Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group Yoga (Experimental): 35 rural teachers in a southwestern Montana school district participating in a trauma-informed yoga intervention
  Interventions: Behavioral: Trauma-Informed Yoga
- No Intervention (No Intervention): No participants were assigned to the No Intervention Arm

INTERVENTIONS:
Behavioral: Trauma-Informed Yoga — 6 weeks of twice weekly trauma-informed yoga for 45 minutes per session
  Arms: Experimental Group Yoga

SUMMARY:
"A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana" is intended to help mitigate stressors that may contribute to poor behavioral and mental health in rural Montana teachers. The immediate goals of this study is to promote student health by supporting teacher wellbeing through a remotely-delivered trauma-informed yoga intervention.

DETAILED DESCRIPTION:
Project Summary: "A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana" is intended to help mitigate stressors that may contribute to poor behavioral and mental health in rural Montana teachers. The immediate goal of this study is to promote student health by supporting teacher wellbeing through a remotely-delivered trauma-informed yoga intervention.

Specific Aim: Expansion of previous pilot study to teachers in the southwestern Montana school district.

Methods: To explore scalability to rural communities without access to yoga instructors, we will implement a limited feasibility study of online yoga delivery to classroom teachers. This study will enroll a minimum 30 Livingston teachers (taught trauma-informed yoga via Zoom), twice weekly for 45-minute trauma-informed yoga sessions during the 6-week intervention period. No participants were assigned to the "No Intervention" arm. To measure physical health outcomes, pre, mid-, and post-intervention cortisol testing will be utilized to evaluate any changes in teacher stress levels before and after the program. Heart rate variability will also be assessed for teachers pre, mid-, and post-intervention using the HeartMath Inner Balance PPG sensor and Em Wave Pro Plus software. To assess behavioral health, pre- and post-survey instruments will collect targeted wellness/mental health data from teachers. An Adverse Childhood Experience Self-Reporting Screener will also be given to participants to establish a baseline of exposure to childhood trauma, which is closely correlated with health outcomes. Teachers will also complete the Teachers' Sense of Self Efficacy Survey and the Professional Quality of Life Index, which are linked to teacher mental health, retention, and career satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Any teacher currently employed by the Livingston school district who wishes to participate in the intervention (up to 35 participants)

Exclusion Criteria:

* Only teachers will be considered for this study (i.e., no school staff, administrators, etc.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Adams, MD, Ph.D, Study Director — Montana State University
Locations (1):
- Park High School, Livingston, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group Yoga: 20 rural teachers in a southwestern Montana school district participating in a trauma-informed yoga intervention
  Trauma-Informed Yoga: 6 weeks of twice weekly trauma-informed yoga for 45 minutes per session
Period: Overall Study
Arm/Group | Experimental Group Yoga
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 20 educators in a rural southwestern Montana school district
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Cortisol Level [Mean (Standard Deviation); unit: micrograms per deciliter] | 0.07 (0.07)

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Cortisol Levels
Description: Participants will provide a saliva sample in which cortisol levels will be analyzed through salivary assay kits (through Salimetrics.com). Samples will be collected on the first day of the intervention, halfway through the intervention, and on the last day of the intervention to determine if the intervention has improved stress levels (as indicated by a reduction in cortisol levels). A biostatistician will provide analysis and conclusion of these samples at the conclusion of the study
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 educators in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
ug/dl
  Pre-Intervention | 0.07 (0.07)
  Post-Intervention | 0.11 (0.08)

2. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: This 9 item questionnaire is designed to evaluate severity of depressive symptoms in participants. It is scored on a Likert scale from 0 (not at all) to 3 (nearly every day) on items linked to depression indicators. The minimum score is a 0 and the maximum score is a 27, and a reduction in score from pre- to post-assessment indicates an improvement in symptomology. Lower scores indicate a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 8.75 (5.674)
  Post-Intervention | 4.85 (3.977)

3. Primary Outcome: Generalized Anxiety Disorder-7 Anxiety Scale (GAD-7)
Description: This 7 item questionnaire is based on a likert scale of 0 (not at all) to 3 (nearly every day) for items related to anxiety disorders. The lowest score is a zero and the maximum score is a 21. A reduction in score from pre- to post-assessment indicates an improvement in symptomology. Lower scores indicate a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 13.9 (6.632)
  Post Intervention | 4.85 (3.99)

4. Primary Outcome: Heart Rate Variability
Description: Participants enrolled will have their heart rate data measured by the HeartMath Institute Inner Balance Bluetooth Sensor and accompanying software for Android or IOS smartphones (Inner Balance) or Inner Balance USB Sensor and accompanying computer software (EmWave Pro Plus (28, 29) The small plastic sensors will clip to the participant's earlobe and send photoplethysmography-derived (PPG) pulse signals via a non-invasive light source and photodetector.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
beats per minute (bpm)
  Pre-Intervention | 1.45 (0.62)
  Post-intervention | 1.45 (0.54)

5. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: The Connor Davidson Resilience Scale (CD-RISC 10) is a unidimensional self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. The minimum value is a 0 and the maximum value is a 100. A higher score indicates higher resilience, which indicates a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 28.35 (6.002)
  Post-intervention | 38.5 (7.119)

6. Secondary Outcome: Professional Quality of Life Index (Pro-QOL)
Description: The Professional Quality of Life Index (Pro-QOL) is self-reporting scale consisting of 30 items measuring levels of compassion satisfaction, secondary trauma, and professional burnout. Respondents rate items on a 5 point Likert scale ranging from 0 (never) to 5 (very often). The minimum score for each subscale is a 10, and the maximum score for each subscale is a 50. Higher scores on compassion satisfaction items indicate higher levels of job enjoyment, whereas higher scores on burnout and secondary trauma items indicate lower levels of job satisfaction. For each of the sub-scales scores are categorized as Low (22 or less), Moderate (between 23 and 41) or High (42 or more). A total sum of each sub-scale is not intended to be measured. Higher scores on the compassion satisfaction scale indicate a better outcome. Lower scores on burnout and secondary trauma indicate a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention Burnout | 34.4 (4.43)
  Post-Intervention Burnout | 23.2 (7.324)
  Pre-Intervention Compassion Satisfaction | 37.95 (7.437)
  Post-Intervention Compassion Satisfaction | 39.2 (6.55)
  Pre-Intervention Secondary Traumatic Stress | 23.9 (8.723)
  Post-Intervention Secondary Traumatic Stress | 22.55 (6.411)

7. Secondary Outcome: Teachers' Sense of Self-Efficacy (Short Form) (TSSE)
Description: The Teachers' Sense of Self-Efficacy is a self-reporting scale consisting of 12 items measuring levels of self-perceived levels of impact on student engagement, instructional strategies, and classroom management. Respondents rate items on a 9 point Likert scale ranging from 1 (nothing) to 9 (a great deal). Higher scores indicate higher self-perceptions of self-efficacy. Higher scores indicate a better outcome. A minimum score isa 12, and a maximum score of 108 is possible on the scale.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 74.85 (20.306)
  Post-Intervention | 82.3 (8.694)

8. Secondary Outcome: PROMIS Sleep Disturbance Scales (PROMIS)
Description: The PROMIS Sleep Disturbance Scale is self-reporting scale consisting of 8 items measuring perceived levels of sleep quality over the previous 7 days. Items are scored on a Likert scale ranging from 1 (not at all) to 5 (very much). Higher scores indicate a greater severity of sleep disturbance. The scale's minimum score is an 8, and the scale's maximum score is 40; therefore, lower scores indicate better quality of sleep. Lower scores indicate a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 23.4 (2.817)
  Post-Intervention | 20.1 (6.456)

9. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a self-reporting scale consisting of 20 items measuring traumatic stress symptoms in the previous month. Items are scored on a Likert scale from 0 (not at all) to 4 (extremely). Higher scores indicate higher levels of traumatic stress in respondents. The scale's minimum score is a zero with a maximum score being an 80. Therefore, lower scores indicate an improvement in traumatic stress symptomology. Lower scores indicate a better outcome.
Time Frame: Pre-Intervention (Baseline), Post-Intervention (Week 6)
Population: 20 rural teachers in a southwestern Montana school district
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group Yoga
Number analyzed (Participants) | 20
score on a scale
  Pre-Intervention | 26 (20.736)
  Post-Intervention | 14.75 (13.436)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: No adverse events occurred.
Arm/Group | Experimental Group Yoga
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05085392/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT05085392/ICF_001.pdf